CLINICAL TRIAL: NCT04312022
Title: Impacts of a Combined Berry Extract Supplement on Endothelial Function, Blood Pressure, Oxygen Utility Capacity, and Fatigue Index in Healthy Young Adults
Brief Title: Impacts of a Combined Berry Extract Supplement on Vascular Function and Oxygen Utility Capacity in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 0436-18-FB
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: anthocyanin; endothelial function; oxygen; vascular function; blood pressure; antioxidant
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover design (1:1)
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor the investigators were aware of the study assignments, which were assigned by a lab member not directly involved in the measurements of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berry extract intake, then Placebo (Experimental): Participants received a single dose of berry extract supplement (hawthorn berry extract, tart cherry extract, and bromelain). After a washout period of 2 weeks, they then received a single dose of the placebo (flour capsule).
  Interventions: Dietary Supplement: Berry extract
- Placebo intake, then Berry extract intake (Placebo Comparator): Participants received a single dose of placebo (flour capsule). After a washout period of 2 weeks, they then received a single dose of berry extract supplement (hawthorn berry extract, tart cherry extract, and bromelain).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Berry extract — Berry extract supplement (hawthorn berry extract, tart cherry extract, bromelain)
  Arms: Berry extract intake, then Placebo
Other: Placebo — Placebo (flour capsule)
  Arms: Placebo intake, then Berry extract intake

SUMMARY:
The purpose of this study is to investigate the impacts of a combined berry extract supplement (hawthorn berry, tart cherry, and bromelain extracts) on total antioxidant capacity, endothelial function, blood pressure, oxygen utility capacity, and fatigue index in healthy young adults.

DETAILED DESCRIPTION:
There are several proposed mechanisms that are thought to contribute to the development of cardiovascular diseases. Although the process is extremely complex, it is well-accepted that elevated levels of reactive oxygen species (ROS) production and inflammation contribute to the systemic vascular dysfunction in cardiovascular diseases. These factors often partially contribute to endothelial dysfunction, elevated blood pressure, reduced oxygen utility capacity, and reduced muscle function. Therefore, by reducing ROS and inflammation, there may be protective effects against vascular dysfunction and thus protection against cardiovascular disease manifestation. Intake of natural anthocyanins and polyphenols derived from fruits and vegetables has been shown to reduce excessive ROS and inflammation in several populations.

Therefore, the purpose of this study was to investigate the impacts of a combined berry extract supplement (hawthorn berry, tart cherry, and bromelain extracts) on total antioxidant capacity, endothelial function, blood pressure, oxygen utility capacity, and fatigue index in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy adult

Exclusion Criteria:

* cardiovascular disease
* neurological disorder
* metabolic disorder
* respiratory disorder
* renal diseases
* musculoskeletal injury
* bleeding disorder
* allergy to fruit
* pregnant/breast feeding
* taking daily medication (prescription or over-the-counter)

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-04 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Song-Young Park, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants completed this study and participated in both arms (berry extract and placebo) in a randomized crossover study design with a 2 wk washout period.
Groups:
- Berry Extract, Then Placebo: Participants first received a single dose of berry extract supplementation (Hawthorn extract 465mg, Tart cherry powder 480mg, and Bromelain 400mg). After a 2 week washout period, they then received a single dose of placebo (tapioca powder).
- Placebo, Then Berry Extract: Participants first received a single dose of placebo (tapioca powder). After a 2 week washout period, they then received a single dose of berry extract supplementation (Hawthorn extract 465mg, Tart cherry powder 480mg, and Bromelain 400mg).
Period: First Intervention (1 Day)
Arm/Group | Berry Extract, Then Placebo | Placebo, Then Berry Extract
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Berry Extract, Then Placebo | Placebo, Then Berry Extract
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Berry Extract, Then Placebo | Placebo, Then Berry Extract
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: n = 18 participants completed the study in a randomized crossover study design
Groups:
- Total: Total of all reporting groups
Arm/Group | Berry Extract, Then Placebo | Placebo, Then Berry Extract | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.2) | 24.2 (4.1) | 24.8 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 6 | 3 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body height [Mean (Standard Deviation); unit: centimeters] | 174.06 (6.1) | 172.4 (7.0) | 173.3 (6.2)
Body mass [Mean (Standard Deviation); unit: kilograms] | 76.7 (9.5) | 76.8 (13.1) | 76.8 (10.8)
Body composition (body fat percentage) [Mean (Standard Deviation); unit: percentage of body fat] | 18.3 (4.4) | 24.1 (5.4) | 21.2 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function
Description: Endothelial function was measured using flow-mediated dilation in percents (%). A higher value represents a better outcome. Scale range for endothelial function is approximately 8-12% for healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percent dilation
Groups:
- Berry Extract Intake: Intake of a berry extract supplement (hawthorn berry extract, tart cherry extract, and bromelain)
  Berry extract: Berry extract supplement (hawthorn berry extract, tart cherry extract, bromelain)
- Placebo Intake: Intake of a placebo (flour capsule)
  Placebo: Placebo (flour capsule)
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
percent dilation | 11.7 (2.9) | 8.2 (3.1)

2. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure was measured as millimeters of mercury (mmHg). Higher values represent a worse outcome. Scale range for systolic blood pressure is approximately 110-129 for most healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
millimeters of mercury | 110.0 (10.0) | 112.5 (10.3)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure was measured as millimeters of mercury (mmHg). Higher values represent a worse outcome. Scale range for systolic blood pressure is approximately 70-79 mmHg for most healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
millimeters of mercury | 72.8 (7.0) | 72.4 (7.4)

4. Secondary Outcome: Oxygen Utility Capacity (Tissue Saturation Index)
Description: Oxygen utility capacity was measured as tissue saturation index in percent (%). Higher values represent a better outcome. Scale range for tissue saturation index (TSI) is approximately 60-90% for most healthy populations at rest.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
percent | 71.5 (10.4) | 64.3 (24.3)

5. Secondary Outcome: Exercise Fatigue Index During Leg Extension
Description: Index of fatigue during leg extension exercise. A lower value represents a better outcome. Scale range is ~15 - 35% for most healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percent fatigue
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
percent fatigue | 27.4 (11.0) | 25.0 (8.6)

6. Secondary Outcome: Exercise Fatigue Index During Leg Flexion
Description: Fatigue index was quantified during isokinetic contraction of the participants dominant leg before and after berry extract and placebo intake using an isokinetic dynamometer. Test consisted of mild resistance at 240°/s to induce and measure muscular fatigue. Fatigue index = (initial peak torque - final peak torque)/initial peak torque x 100). A lower value represents a better outcome. Scale range is ~15 - 35% for most healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percent fatigue
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
percent fatigue | 24.9 (11.2) | 24.8 (11.8)

7. Secondary Outcome: Plasma Total Antioxidant Capacity
Description: Total antioxidant capacity assessed from the venous blood (plasma). A higher value represents a better outcome. Scale range is 10 - 20 millimoles per milliliter for most healthy populations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: millimoles per milliliter
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
millimoles per milliliter | 15.8 (9.0) | 15.0 (8.5)

8. Secondary Outcome: Oxygenated Hemoglobin
Description: Oxygenated hemoglobin was measured in arbitrary units (a.u.). Higher values represent a better outcome. Scale range for oxygenated hemoglobin is ~5-15 a.u. in healthy populations
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: arbitrary units (a.u.)
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
arbitrary units (a.u.) | 10.1 (7.1) | 9.6 (8.1)

9. Secondary Outcome: Deoxygenated Hemoglobin
Description: Deoxygenated hemoglobin was measured in arbitrary units (a.u.). Lower values represent a better outcome. Scale range for deoxygenated hemoglobin is ~ - 5-5 in healthy populations
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: arbitrary units (a.u.)
Arm/Group | Berry Extract Intake | Placebo Intake
Number analyzed (Participants) | 18 | 18
arbitrary units (a.u.) | -0.4 (1.3) | -2.7 (8.7)

ADVERSE EVENTS:
Time Frame: 2 wk
Arm/Group | Berry Extract Intake | Placebo Intake
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04312022/Prot_SAP_000.pdf